CLINICAL TRIAL: NCT05358860
Title: Safety and Efficacy of Sofwave Treatment for Acne Scars Appearance Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sofwave09
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
Keywords: Acne Scars
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Acne Scars (Experimental)
  Interventions: Device: Sofwave

INTERVENTIONS:
Device: Sofwave — The Sofwave System, comprised of an applicator and a console, generates high intensity, non-focused ultrasonic energy which can be delivered percutaneously to tissues.
  Other Names: SUPERB

SUMMARY:
Open-label, non-randomized, prospective, multi-center, self-controlled clinical study with masked evaluation.

DETAILED DESCRIPTION:
Eligible patients will receive 3 treatments (4-6 weeks apart) on the facial acne scars using Sofwave System.

Treatment may be administered after the enrollment and screening at the first visit, or it may occur later following the enrollment and screening activities based on site scheduling availabilities.

All patients will return to the clinic for one follow up visit at 3 months ± 3 weeks post last treatment (FU1). Methodology described in the protocol to evaluate efficacy and safety of treatments will be carried out at each visit at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects > 22 years of age and < 80 years of age.
2. For female subjects, not pregnant or lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide) or abstinence.
3. Seeking treatment for facial acne scars.
4. Have visible mild to moderate facial acne scars.
5. Agree not to undergo any other facial acne scars treatments for a period of 3 months following Sofwave treatments.
6. Willing to have photographs of the treated areas. Agree for de-identified study images to be used in evaluations, publications and presentations.
7. Able and willing to comply with all visits, treatments and evaluations schedules and requirements.
8. Able to understand and provide written Informed Consent

Exclusion Criteria:

1. Pregnant or planning to become pregnant during the duration of the study, having given birth less than 3 months ago, and/or breast feeding
2. Current smoker or has history of heavy smoking (25 cigarettes per day or more) in past 10 years.
3. History of severe migraine tendency.
4. History of Epileptic seizures.
5. History of chronic drug or alcohol abuse.
6. Taking Isotretinoin or other oral retinoid within the past 6 months; taking anti-platelet or anti-coagulant within the past 2 weeks.
7. Medical disorder that may hinder the wound healing or immune response (such as blood disorder, inflammatory disease, etc.)
8. Presence of a metal stent or implant in the facial area.
9. Known allergy to tetracaine, Xylocaine or epinephrine.
10. Active malignancy or history of malignancy in the past 5 years.
11. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders (i.e. any disease state that in the opinion of the investigator may interfere with the anesthesia, treatment, or healing process).
12. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
13. Presence of any active systemic or local infections.
14. Severe or cystic facial acne, acutance uses during past 6 months.
15. History of cosmetic treatments in the facial area to be treated, including facial skin-tightening procedure within the 6 months; injectable (Botox or fillers of any type) within the 6 months; ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep facial peels within the past 12 months; facelift or blepharoplasty within the past 12 months.
16. Inability to understand the protocol or to give informed consent
17. On-going use of psychiatric medication
18. Unable or unwilling to comply with the study requirements and procedures
19. Currently enrolled in a clinical study of any other unapproved investigational drug or device
20. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of change of acne scars appearance, as assessed by independent masked evaluators at 3 months post last treatment session. | 1 year
  following Sofwave treatments based on 6 points simplified Acne Severity Scale (ASS), as evaluated by independent masked reviewers.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - SLSS, a Division of Schweiger Dermatology Group Research Office, Hackensack, New Jersey
  - UnionDerm, New York, New York
  - Laser & Skin Surgery Center of New York®, New York, New York
  - New York Laser & Skin Care, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided